CLINICAL TRIAL: NCT03792191
Title: Ultrasonography Versus Palpation for Spinal Anesthesia in Obese Parturients Undergoing Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Mohamed Tawfik, Lecturer, Department of anesthesia and surgical intensive care, Primary investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD.18.02.29
Record Dates: First submitted 2019-01-01; First posted 2019-01-03 (Actual); Results first posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Anesthesia, Spinal; Cesarean Section; Spinal Ultrasound
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasonography (Experimental): Preprocedural lumbar spinal ultrasonography and skin marking. Spinal anesthesia will be administered with injection of intrathecal bupivacaine and intrathecal fentanyl.
  Interventions: Radiation: Lumbar Spinal Ultrasonography; Procedure: Spinal Anesthesia; Drug: Intrathecal Bupivacaine; Drug: Intrathecal Fentanyl
- Palpation (Active Comparator): Sham ultrasound procedure. Conventional landmark palpation and skin marking.Spinal anesthesia will be administered with injection of intrathecal bupivacaine and intrathecal fentanyl.
  Interventions: Radiation: Sham Ultrasound Procedure; Procedure: Conventional Landmark Palpation; Procedure: Spinal Anesthesia; Drug: Intrathecal Bupivacaine; Drug: Intrathecal Fentanyl

INTERVENTIONS:
Radiation: Lumbar Spinal Ultrasonography — Ultrasonography of the lumbar spines using an 8-2 MHz curved array transducer. Identification of the intervertebral space with the best image. Marking the patient's skin with horizontal and vertical lines over the L3-L4 and L2-L3 intervertebral spaces.
  Arms: Ultrasonography
Radiation: Sham Ultrasound Procedure — Moving the ultrasound probe on the patient's back with the machine in the freeze position.
  Arms: Palpation
Procedure: Conventional Landmark Palpation — Conventional palpation of the anatomical landmarks. The line crossing the iliac crests (Tuffier line) is assumed to cross the spine at L4 spinous process or L3-L4 intervertebral space. Identification of the widest intervertebral space. Marking the patient's skin with horizontal and vertical lines over the L3-L4 and L2-L3 intervertebral spaces.
  Arms: Palpation
Procedure: Spinal Anesthesia — Spinal anesthesia using a 25- or 22-gauge spinal needle
Drug: Intrathecal Bupivacaine — Bupivacaine 12.5 mg (2.5 mL 0.5%) will be administered in the subarachnoid space
Drug: Intrathecal Fentanyl — Fentanyl 15 μg will be administered in the subarachnoid space

SUMMARY:
The study will compare between preprocedural ultrasonography and the conventional palpation technique for spinal anesthesia in obese parturients undergoing elective cesarean delivery

DETAILED DESCRIPTION:
This randomized, controlled, double-blind study will be conducted on ASA physical status II-III obese parturients with full-term singleton pregnancy undergoing elective cesarean delivery under spinal anesthesia. The study subjects will be assigned to 2 equal groups. In the ultrasonography group, lumbar spinal ultrasonography will be performed before administration of spinal anesthesia. In the palpation group, conventional palpation of the anatomical landmarks will be performed.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status II-III parturients
* Full term singleton pregnancy
* Body mass index ≥ 35 Kg/m2

Exclusion Criteria:

* Age < 19 years
* Women presenting in labor
* Contraindications to neuraxial anesthesia (Coagulopathy, increased intracranial pressure, or local skin infection)
* Significant spinal deformities or previous spinal surgery
* Preeclampsia

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Tawfik, MD, Study Director — Mansoura University Hospital; Mohamed A Tolba, MSc, Principal Investigator — Mansoura University Hospital
Locations (1):
- Department of Anesthesia, Mansoura University Hospitals, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tawfik MM, Tolba MA, Ismail OM, Messeha MM. Ultrasonography versus palpation for spinal anesthesia in obese parturients undergoing cesarean delivery: a randomized controlled trial. Reg Anesth Pain Med. 2024 Jan 11;49(1):41-48. doi: 10.1136/rapm-2022-104272. PMID 37188389

RESULTS

PARTICIPANT FLOW:
Groups:
- Ultrasonography: Preprocedural lumbar spinal ultrasonography and skin marking. Spinal anesthesia was administered with injection of intrathecal bupivacaine and intrathecal fentanyl.
  Lumbar Spinal Ultrasonography: Ultrasonography of the lumbar spines using an 8-2 MHz curved array transducer. Identification of the interspace with the best image. Marking the patient's skin with horizontal and vertical lines over the L3-L4 and L2-L3 interspaces.
  Spinal Anesthesia: Spinal anesthesia using a 25- or 22-gauge spinal needle
  Intrathecal Bupivacaine: Bupivacaine 12.5 mg (2.5 mL 0.5%) was administered in the subarachnoid space
  Intrathecal Fentanyl: Fentanyl 15 μg was administered in the subarachnoid space
- Palpation: Sham ultrasound procedure. Conventional landmark palpation and skin marking. Spinal anesthesia was administered with injection of intrathecal bupivacaine and intrathecal fentanyl.
  Sham Ultrasound Procedure: Sliding the ultrasound probe on the patient's back with the machine in the freeze position.
  Conventional Landmark Palpation: Conventional palpation of the anatomical landmarks. The line crossing the iliac crests (Tuffier line) was assumed to cross the spine at L4 spinous process or L3-L4 intervertebral space. Identification of the widest interspace. Marking the patient's skin with horizontal and vertical lines over the L3-L4 and L2-L3 interspaces.
  Spinal Anesthesia: Spinal anesthesia using a 25- or 22-gauge spinal needle
  Intrathecal Bupivacaine: Bupivacaine 12.5 mg (2.5 mL 0.5%) was administered in the subarachnoid space
  Intrathecal Fentanyl: Fentanyl 15 μg was administered in the subarachnoid space
Period: Overall Study
Arm/Group | Ultrasonography | Palpation
Started | 140 | 140
Completed | 140 | 140
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultrasonography | Palpation | Total
Number analyzed (Participants) | 140 | 140 | 280
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.2 (5.9) | 30.3 (5.5) | 30.3 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 140 | 280
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Egypt | 140 | 140 | 280
Height [Mean (Standard Deviation); unit: cm] | 159.5 (6.1) | 160 (6.1) | 159.7 (6.1)
Weight [Median (Full Range); unit: kg] | 102 [80 to 160] | 103 [76 to 140] | 102 [76 to 160]
Body mass index [Median (Full Range); unit: kg/m^2] | 40.2 [35.2 to 61] | 39.2 [35 to 58.3] | 39.8 [35 to 61]
Gestational age (weeks) [Median (Full Range); unit: weeks] | 38 [37 to 41] | 38 [37 to 40] | 38 [37 to 41]
Nulliparous [Count of Participants; unit: Participants] | 21 | 19 | 40
Ease of landmark palpation [Count of Participants; unit: Participants] — A 4-point scale (1 = the spinous processes and the interspaces can be identified by light palpation; 2 = the spinous processes and the interspaces can be identified by deep palpation; 3 = the spinous processes only can be identified by deep palpation, and the interspaces cannot be identified; 4 = neither the spinous processes nor the interspaces can be identified).
  Participants
    1 | 11 | 17 | 28
    2 | 57 | 62 | 119
    3 | 63 | 54 | 117
    4 | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Needle Passes Required to Obtain Free Cerebrospinal Fluid Flow
Description: Needle pass is any forward introduction of the spinal needle after its complete or incomplete withdrawal, including the first attempt.
Time Frame: Assessed from starting the first attempt of spinal anesthesia until successful administration of spinal anesthesia, an average of 10 minutes
Measure: Median (Full Range); unit: needle passes
Groups:
- Palpation: Sham ultrasound procedure. Conventional landmark palpation and skin marking. Spinal anesthesia was administered with injection of intrathecal bupivacaine and intrathecal fentanyl.
  Sham Ultrasound Procedure: Moving the ultrasound probe on the patient's back with the machine in the freeze position.
  Conventional Landmark Palpation: Conventional palpation of the anatomical landmarks. The line crossing the iliac crests (Tuffier line) was assumed to cross the spine at L4 spinous process or L3-L4 intervertebral space. Identification of the widest interspace. Marking the patient's skin with horizontal and vertical lines over the L3-L4 and L2-L3 interspaces.
  Spinal Anesthesia: Spinal anesthesia using a 25- or 22-gauge spinal needle
  Intrathecal Bupivacaine: Bupivacaine 12.5 mg (2.5 mL 0.5%) was administered in the subarachnoid space
  Intrathecal Fentanyl: Fentanyl 15 μg was administered in the subarachnoid space
Arm/Group | Ultrasonography | Palpation
Number analyzed (Participants) | 140 | 140
needle passes | 3 [1 to 34] | 3 [1 to 23]
Statistical Analysis 1: Comparison: Ultrasonography vs Palpation; Test type: Superiority; p = 0.62, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.00007, 95% CI 2-sided [-0.00005 to 1]

2. Secondary Outcome: Number of Skin Punctures Required to Obtain Free Cerebrospinal Fluid Flow
Description: Skin puncture is any separate skin puncture by the spinal needle after its complete withdrawal, including the first attempt.
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: skin punctures
Arm/Group | Ultrasonography | Palpation
Number analyzed (Participants) | 140 | 140
skin punctures | 1 [1 to 6] | 1 [1 to 4]
Statistical Analysis 1: Comparison: Ultrasonography vs Palpation; Test type: Superiority; p = 0.58, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Rate of Successful Obtaining of Free Cerebrospinal Fluid Flow at the First Needle Pass
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasonography | Palpation
Number analyzed (Participants) | 140 | 140
Participants | 40 | 45
Statistical Analysis 1: Comparison: Ultrasonography vs Palpation; Test type: Superiority; p = 0.6, Chi-squared, Corrected; Risk Difference (RD) = -0.036, 95% CI 2-sided [-0.15 to 0.079]

4. Secondary Outcome: Rate of Successful Obtaining of Free Cerebrospinal Fluid Flow at the First Skin Puncture
Description: as for outcome 2
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasonography | Palpation
Number analyzed (Participants) | 140 | 140
Participants | 108 | 111
Statistical Analysis 1: Comparison: Ultrasonography vs Palpation; Test type: Superiority; p = 0.77, Chi-squared, Corrected; Risk Difference (RD) = -0.021, 95% CI 2-sided [-0.125 to 0.082]

5. Secondary Outcome: Duration of the Spinal Procedure
Description: The duration from starting the first skin puncture by the spinal needle to obtaining free CSF flow
Time Frame: Assessed from enrollment in the study until completion of cesarean delivery
Measure: Median (Full Range); unit: seconds
Arm/Group | Ultrasonography | Palpation
Number analyzed (Participants) | 140 | 140
seconds | 76 [26 to 734] | 59 [19 to 700]
Statistical Analysis 1: Comparison: Ultrasonography vs Palpation; Test type: Superiority; p = 0.077, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 8, 95% CI 2-sided [-1 to 20]

6. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction from the procedure assessed immediately after intrathecal injection using a 5-point scale (1 = very unsatisfied; 2 = unsatisfied; 3 = fair; 4 = satisfied; and 5 = very satisfied).
Time Frame: Assessed at 1 minute after intrathecal injection
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Ultrasonography | Palpation
Number analyzed (Participants) | 140 | 140
units on a scale | 5 [1 to 5] | 4 [1 to 5]
Statistical Analysis 1: Comparison: Ultrasonography vs Palpation; Test type: Superiority; p = 0.1, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.00003, 95% CI 2-sided [-0.00001 to 0.00003]

7. Secondary Outcome: Number of Participants With Vascular Puncture
Description: Number of participants with unintentional vascular puncture by the needle during performing the spinal procedure
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasonography | Palpation
Number analyzed (Participants) | 140 | 140
Participants | 9 | 9
Statistical Analysis 1: Comparison: Ultrasonography vs Palpation; Test type: Superiority; p > 0.99, Chi-squared, Corrected

8. Secondary Outcome: Number of Participants With Paresthesia
Description: Number of participants with paresthesia reported by the subjects during performing the spinal procedure
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasonography | Palpation
Number analyzed (Participants) | 140 | 140
Participants | 16 | 17
Statistical Analysis 1: Comparison: Ultrasonography vs Palpation; Test type: Superiority; p > 0.99, Chi-squared, Corrected

9. Secondary Outcome: Number of Participants With Failure to Obtain Free Cerebrospinal Fluid Flow
Description: Number of participants with failure to obtain free cerebrospinal fluid flow after adequate needle passes at 6 separate skin punctures.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasonography | Palpation
Number analyzed (Participants) | 140 | 140
Participants | 0 | 0

10. Secondary Outcome: Number of Participants With Failed Spinal Block
Description: Number of participants with failed spinal block defined as an upper sensory level below T6 assessed by pinprick.
Time Frame: Assessed up to 20 minutes after intrathecal injection
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasonography | Palpation
Number analyzed (Participants) | 140 | 140
Participants | 3 | 4
Statistical Analysis 1: Comparison: Ultrasonography vs Palpation; Test type: Superiority; p > 0.99, Fisher Exact

ADVERSE EVENTS:
Time Frame: From enrollment in the study until home discharge, up to 48 hours
Arm/Group | Ultrasonography | Palpation
All-Cause Mortality (participants affected / at risk) | 0/140 | 0/140
Serious Adverse Events (participants affected / at risk) | 0/140 | 0/140
Other Adverse Events (participants affected / at risk) | 0/140 | 0/140

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-31): https://cdn.clinicaltrials.gov/large-docs/91/NCT03792191/Prot_SAP_000.pdf